CLINICAL TRIAL: NCT02554721
Title: Effect of Cilostazol as an add-on Treatment to a Single Antiplatelet Agent (Acetylsalicylic Acid or Clopidogrel) on Platelet Function Testing and Bleeding Time in Healthy Volunteers
Brief Title: Pharmacodynamic Study of Cilostazol in Healthy Volunteers
Acronym: CiloMecT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-13-102; 2013-002633-38 (EudraCT Number)
Record Dates: First submitted 2015-09-15; First posted 2015-09-18 (Estimated); Results first posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Healthy
Keywords: Healthy Volunteers
MeSH Terms: interventions — Cilostazol; Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (CYP2C19 Wild Type) (Experimental): Trial period A: Cilostazol 100 mg twice daily for 1 week (Days 1-7) Trial period B: Wash out period (Days 8-14) Trial period C: Acetylsalicylic acid 100 mg once daily for 1 week (Days 15-21) Trial period D: Cilostazol 100 mg twice daily and Acetylsalicylic acid 100mg once daily for 1 week (Days 22-28)
  Interventions: Drug: Cilostazol; Drug: Acetylsalicylic acid
- Group 2 (CYP2C19 Wild Type) (Experimental): Trial period A: Cilostazol 100 mg twice daily for 1 week (Days 1-7) Trial period B: Wash out period (Days 8-14) Trial period C: Clopidogrel 75 mg once daily for 1 week (Days 15-21) Trial period D: Cilostazol 100 mg twice daily and Clopidogrel 75 mg once daily for 1 week (Days 22-28)
  Interventions: Drug: Cilostazol; Drug: Clopidogrel
- Group 3 (CYP2C19 heterozygous (*1/*2) ) (Experimental): Trial period A: Cilostazol 100 mg twice daily for 1 week (Days 1-7) Trial period B: Wash out period (Days 8-14) Trial period C: Clopidogrel 75 mg once daily for 1 week (Days 15-21) Trial period D: Cilostazol 100 mg twice daily and Clopidogrel 75 mg once daily for 1 week (Days 22-28)
  Interventions: Drug: Cilostazol; Drug: Clopidogrel
- Group 4 (CYP2C19 homozygous (*2/*2)) (Experimental): Trial period A: Cilostazol 100 mg twice daily for 1 week (Days 1-7) Trial period B: Wash out period (Days 8-14) Trial period C: Clopidogrel 75 mg once daily for 1 week (Days 15-21) Trial period D: Cilostazol 100 mg twice daily and Clopidogrel 75 mg once daily for 1 week (Days 22-28)
  Interventions: Drug: Cilostazol; Drug: Clopidogrel

INTERVENTIONS:
Drug: Cilostazol
Drug: Acetylsalicylic acid
  Arms: Group 1 (CYP2C19 Wild Type)
Drug: Clopidogrel
  Arms: Group 2 (CYP2C19 Wild Type); Group 3 (CYP2C19 heterozygous (*1/*2) ); Group 4 (CYP2C19 homozygous (*2/*2))

SUMMARY:
The primary objective of this study is to investigate the effects of Cilostazol, Acetylsalycylic acid and Clopidogrel alone as well as combinations of Cilostazol/Acetylsalicylic acid and Cilostazol/ Clopidogrel on ex-vivo Platelet Function (PF) testing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian male subjects
* Able to read, to write and to fully understand German language
* Provision of written informed consent before screening and baseline
* BMI between 19.0 and 30.0 kg/m2, inclusive and body weight between 50.0 and 100.0 kg, inclusive
* Good general health as determined by the investigator by medical history, physical examination, vital signs, electrocardiogram, baseline and safety lab

Exclusion Criteria:

* Personal or family history of bleeding disorders, or reasonable suspicion of vascular malformations, including aneurysms
* Known predisposition to bleeding (e.g. active peptic ulceration, recent (within 6 month) haemorrhagic stroke, proliferative diabetic retinopathy, poorly controlled hypertension)
* Use of antibiotics within thirty (30) days prior to screening and until baseline visit
* Clinically significant abnormalities in medical history, physical examination, vital signs, electrocardiogram, baseline and safety lab
* Supine pulse rate > 100 beats/min or <50 beats/min
* Systolic blood pressure <100 or >140 mmHg
* Diastolic blood pressure <50 or >90 mmHg
* Concomitant use of any other medication including over-the-counter preparations

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Osamu Sato, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Bad Krozingen, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 77 healthy adult male participants were enrolled. Following administration of cilostazol in Period A and wash-out in Period B, participants were stratified according to CYP2C19 genotype and assigned to Groups 1-4 for further treatment in Periods C and D. Two participants who received cilostazol in Period A were not assigned to a group.
Groups:
- Group 1 (CYP2C19 EM): Participants received cilostazol 100 milligrams (mg) twice daily (BID) for 7 consecutive days from Day 1 to Day 7 (Period A). A 7-day wash-out period (Period B) allowed a return to baseline in relation to platelet function (PF) and skin bleeding time (BT) from Day 8 to Day 14. Participants who failed to return to baseline with respect to PF and skin BT were retested within a further week (Day 15 to Day 21). Participants with normal, extensive metabolic (EM) activity (CYP2C19 EM) received ASA 100 mg once daily (QD) for 7 consecutive days from Day 15 to Day 21 or Day 22 to Day 28 for participants who failed to return to baseline with respect to PF testing and skin BT at the scheduled visit 7 days after last administration of cilostazol (from Day 1 to Day 7) (Period C). In the following week, participants received cilostazol 100 mg BID as an add-on therapy to ASA 100 mg QD for 7 consecutive days from Day 22 to Day 28 or Day 29 to Day 35 (Period D).
- Group 2 (CYP2C19 EM): Participants received cilostazol 100 mg BID for 7 consecutive days from Day 1 to Day 7 (Period A). A 7- day wash-out period (Period B) allowed a return to baseline in relation to PF and skin BT from Day 8 to Day 14. Participants who failed to return to baseline with respect to PF and skin BT were retested within a further week (Day 15 to Day 21). Participants with normal EM activity (CYP2C19 EM) received clopidogrel 75 mg QD for 7 consecutive days from Day 15 to Day 21 or Day 22 to Day 28 for participants who failed to return to baseline with respect to PF testing and skin BT at the scheduled visit 7 days after last administration of cilostazol (from Day 1 to Day 7) (Period C). In the following week, participants received cilostazol 100 mg BID as an add-on therapy to clopidogrel 75 mg QD for 7 consecutive days from Day 22 to Day 28 or Day 29 to Day 35 (Period D).
- Group 3 (CYP2C19 IM): Participants received cilostazol 100 mg BID for 7 consecutive days from Day 1 to Day 7 (Period A). A 7- day wash-out period (Period B) allowed a return to baseline in relation to PF and skin BT from Day 8 to Day 14. Participants who failed to return to baseline with respect to PF and skin BT were retested within a further week (Day 15 to Day 21). Participants with intermediate metabolic (IM) activity (CYP2C19 IM) received clopidogrel 75 mg QD for 7 consecutive days from Day 15 to Day 21 or Day 22 to Day 28 for participants who failed to return to baseline with respect to PF testing and skin BT at the scheduled visit 7 days after last administration of cilostazol (from Day 1 to Day 7) (Period C). In the following week, participants received cilostazol 100 mg BID as an add-on therapy to clopidogrel 75 mg QD for 7 consecutive days from Day 22 to Day 28 or Day 29 to Day 35 (Period D).
- Group 4 CYP2C19 PM): Participants received cilostazol 100 mg BID for 7 consecutive days from Day 1 to Day 7 (Period A). A 7- day wash-out period (Period B) allowed a return to baseline in relation to PF and skin BT from Day 8 to Day 14. Participants who failed to return to baseline with respect to PF and skin BT were retested within a further week (Day 15 to Day 21). Participants with poor metabolic (PM) activity (CYP2C19 PM) received clopidogrel 75 mg QD for 7 consecutive days from Day 15 to Day 21 or Day 22 to Day 28 for participants who failed to return to baseline with respect to PF testing and skin BT at the scheduled visit 7 days after last administration of cilostazol (from Day 1 to Day 7) (Period C). In the following week, participants received cilostazol 100 mg BID as an add-on therapy to clopidogrel 75 mg QD for 7 consecutive days from Day 22 to Day 28 or Day 29 to Day 35 (Period D).
- Not Assigned: Two participants who received cilostazol in Period A were not assigned to a group.
Period: Overall Study
Arm/Group | Group 1 (CYP2C19 EM) | Group 2 (CYP2C19 EM) | Group 3 (CYP2C19 IM) | Group 4 CYP2C19 PM) | Not Assigned
Started | 20 | 19 | 19 | 17 | 2
Completed | 19 | 19 | 19 | 17 | 0
Not Completed | 1 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 1
Not completed — Noncompliance | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All subjects who received at least 1 dose of trial medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (CYP2C19 EM) | Group 2 (CYP2C19 EM) | Group 3 (CYP2C19 IM) | Group 4 CYP2C19 PM) | Not Assigned | Total
Number analyzed (Participants) | 20 | 19 | 19 | 17 | 2 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.8 (4.3) | 28.3 (6.5) | 25.9 (4.6) | 24.2 (4.0) | 26.5 (4.9) | 26.1 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 20 | 19 | 19 | 17 | 2 | 77
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 20 | 19 | 19 | 17 | 2 | 77
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 20 | 19 | 19 | 17 | 2 | 77

OUTCOME MEASURES:

1. Primary Outcome: Ex-vivo Inhibition Of Platelet Aggregation (IPA)
Description: The effect of ASA in combination with cilostazol and clopidogrel in combination with cilostazol on IPA was determined ex vivo in citrated platelet rich plasma (PRP) after stimulation of aggregation by low-level adenosine diphosphate (ADP) (5 micromolar [uM]) and arachidonic acid (AA) (500 milligrams/liter [mg/L]). Light transmission aggregometry (LTA) was used to measure residual aggregation (the percentage of aggregation 5 minutes after the addition of ADP or AA). Results are reported as the 95% confidence intervals for the reported geometric mean ratios (GMRs) ([cilostazol+reference (ASA or clopidogrel)]/reference) for IPA.
Time Frame: Baseline, Visit 5 (Day 22-29)
Population: Full Analysis Set: All subjects who completed both periods of treatment with reference medication alone (Period C) and treatment with reference medication and cilostazol (Period D)
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Groups:
- Acetylsalicylic Acid - Cilostazol: Participants with normal CYP2C19 activity (EM) (Group 1) who received ASA 100 mg QD for 7 consecutive days from Day 15 to Day 21 (Period C) went on to receive cilostazol 100 mg BID as an add-on therapy to ASA 100 mg QD for 7 consecutive days from Day 22 to Day 28 or Day 29 to Day 35 (Period D).
- Clopidogrel - Cilostazol: Participants with EM, IM, and PM CYP2C19 activity (Groups 2-4, respectively) who received clopidogrel 75 mg QD for 7 consecutive days from Day 15 to Day 21 (Period C) went on to receive cilostazol 100 mg BID as an add-on therapy to clopidogrel 75 mg QD for 7 consecutive days from Day 22 to Day 28 or Day 29 to Day 35 (Period D).
Arm/Group | Acetylsalicylic Acid - Cilostazol | Clopidogrel - Cilostazol
Number analyzed (Participants) | 15 | 51
ratio
  5 µM ADP | 0.82 [0.5 to 1.37] | 1.21 [1.09 to 1.35]
  500 mg/L AA | 1.03 [1.01 to 1.05] | 4.42 [3.42 to 5.73]

2. Secondary Outcome: Effects On Skin Bleeding Time (BT)
Description: The effect of ASA in combination with cilostazol and clopidogrel in combination with cilostazol on skin BT (minutes) was determined with the Ivy method, utilizing standardized bleeding with the Surgicutt device. Results include the 95% confidence intervals for the reported GMRs ([cilostazol+reference]/reference) for skin BT.
Time Frame: Visit 5 (Day 22-29)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Acetylsalicylic Acid - Cilostazol | Clopidogrel - Cilostazol
Number analyzed (Participants) | 17 | 51
ratio | 1.31 [1.05 to 1.63] | 1.27 [1.09 to 1.48]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from Day 1 to Day 29
Description: Subjects receiving at least 1 dose of study medication were included in the safety analysis.
Groups:
- Cilostazol: All 77 enrolled participants received cilostazol 100 milligrams (mg) twice daily (BID) for 7 consecutive days from Day 1 to Day 7. A 7-day wash-out period (Period B) allowed a return to baseline in relation to platelet function (PF) and skin bleeding time (BT) from Day 8 to Day 14. Participants who failed to return to baseline with respect to PF and skin BT were retested within a further week (Day 15 to Day 21). After returning to baseline, all participants were stratified and randomized to the following 4 treatment groups in a 1:1:1:1 ratio for treatment in Periods C and D: Group 1, normal, extensive metabolizer (EM); Group 2, EM; Group 3, intermediate metabolizer (IM); Group 4, poor metabolizer (PM).
- Acetylsalicylic Acid: Participants with extensive CYP2C19 activity (EM) received ASA 100 mg QD for 7 consecutive days from Day 15 to Day 21, or Day 22 to Day 28 for participants who failed to return to baseline with respect to PF testing and skin BT at the scheduled visit at 7 days after last administration of cilostazol (from Day 1 to Day 7).
- Clopidogrel: Participants with EM, IM, and PM CYP2C19 activity received clopidogrel 75 mg QD for 7 consecutive days from Day 15 to Day 21, or Day 22 to Day 28 for participants who failed to return to baseline with respect to PF testing and skin BT at the scheduled visit at 7 days after last administration of cilostazol (from Day 1 to Day 7).
- Acetylsalicylic Acid - Cilostazol: Participants with extensive CYP2C19 activity (EM) received cilostazol 100 mg BID as an add-on therapy to ASA 100 mg QD for 7 consecutive days from Day 22 to Day 28 or Day 29 to Day 35.
- Clopidogrel - Cilostazol: Participants with EM, IM, and PM CYP2C19 activity received cilostazol 100 mg BID as an add-on therapy to clopidogrel 75 mg QD for 7 consecutive days from Day 22 to Day 28 or Day 29 to Day 35.
Arm/Group | Cilostazol | Acetylsalicylic Acid | Clopidogrel | Acetylsalicylic Acid - Cilostazol | Clopidogrel - Cilostazol
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/20 | 0/55 | 0/20 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/20 | 0/55 | 0/20 | 0/55
Other Adverse Events (participants affected / at risk) | 62/77 | 3/20 | 3/55 | 10/20 | 41/55
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cilostazol (N=77) | Acetylsalicylic Acid (N=20) | Clopidogrel (N=55) | Acetylsalicylic Acid - Cilostazol (N=20) | Clopidogrel - Cilostazol (N=55)
Palpitations (Cardiac disorders) | 5 | 0 | 0 | 2 | 3
Headache (Nervous system disorders) | 60 | 1 | 2 | 10 | 38
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 1 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-03-07): https://cdn.clinicaltrials.gov/large-docs/21/NCT02554721/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/21/NCT02554721/SAP_001.pdf